CLINICAL TRIAL: NCT06305195
Title: Potential Correlation Between Heart Rate Variability With Cardiovascular Risk at Different Stages of Metabolic Syndrome: Impact of Some Antidiabetic Drugs
Brief Title: Potential Correlation Between Heart Rate Variability With Cardiovascular Risk at Different Stages of Metabolic Syndrome
Status: Recruiting | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Hala Abo El Hassan, Teacher assistant, Alexandria University
Other Study IDs: 0107766
Record Dates: First submitted 2024-02-11; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-diabetic individuals: adults (18-70 Years) with glycated hemoglobin (HBA1C) <5.7 and/or Fasting blood glucose <100 mg/L and with no classic symptoms of hyperglycemia
  Interventions: Diagnostic Test: heart rate variability test
- Pre-diabetic:: adults (18-70 Years) who fulfil one of the American Diabetes Association (ADA) criteria :
  * glycated hemoglobin (HBA1C) =5.7-6.4%
  * Fasting blood glucose 100 mg/dL to 125 mg/dL. Fasting is deﬁned as no caloric intake for at least 8 hours.
  Interventions: Diagnostic Test: heart rate variability test
- Diabetic patients :: adults (18-70 Years) who fulfil one of the American Diabetes Association (ADA) criteria:
  * glycated hemoglobin (HBA1C) ≥6.5%
  * Fasting blood glucose ≥126 mg/dL.
  * A random plasma glucose ≥200 mg/dL. Random is any time of the day without regard to the meals.
  Interventions: Diagnostic Test: heart rate variability test

INTERVENTIONS:
Diagnostic Test: heart rate variability test — First, the patient is required to lie on their back to have a 5-minute continuous ECG recorded, without performing any maneuvers.
  Following this, deep breath test, Valsalva and stand test are performed.
  Other Names: Cardiac autonomic reflex tests (CARTs); blood tests

SUMMARY:
The study aims to assess the beat-to-beat Heart rate variability (HRV) in different stages of metabolic diseases, including pre-diabetic and diabetic patients, compared to non-diabetic individuals.

Heart rate variability will be compared for some antidiabetic drugs used in different stages of metabolic diseases and correlated to different metabolic and inflammatory mediators.

ELIGIBILITY:
Inclusion Criteria:

1. Non-diabetic individuals: adults (18-70 Years) with glycated hemoglobin (HBA1C)<5.7 and/or Fasting blood glucose <100 mg/L and with no classic symptoms of hyperglycemia
2. Pre-diabetic: adults (18-70 Years) who fulfil one of the American Diabetes Association (ADA) criteria :

   * glycated hemoglobin (HBA1C) =5.7-6.4%
   * Fasting blood glucose level = 100 mg/dL to 125 mg/dL. Fasting is deﬁned as no caloric intake for at least 8 hours.
3. Diabetic patients: adults (18-70 Years) who fulfil one of the American Diabetes Association (ADA) criteria:

   * glycated hemoglobin (HBA1C) ≥6.5%
   * Fasting blood glucose ≥126 mg/dL.
   * A random plasma glucose ≥200 mg/dL. Random is any time of the day without regard to the meals.

Exclusion Criteria:

* Pediatric and elderly subjects
* Pregnant subjects
* Those with active Myocardial infarction
* Those with acute decompensated heart failure
* Patients with pacemaker
* Patients with persistent Atrial fibrillation, long-standing persistent and permanent Atrial fibrillation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients aged 18-70 Years either diabetic, pre-diabetic or non-diabetic should not have one of the following criteria:
  * Pediatric and elderly subjects
  * Pregnant subjects
  * Those with active Myocardial infarction
  * Those with acute decompensated heart failure
  * Patients with pacemaker
  * Patients with persistent Atrial fibrillation, long-standing persistent and permanent Atrial fibrillation
  * Amputated patients
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
Beat-to-beat Heart rate variability | one year
  •It will be measured Different stages of metabolic diseases among non-diabetic, diabetic and prediabetic subjects
body mass index | one year
  Measuring body weight in kilograms (kg) and height in centimeters (cm) to calculate the Body Mass Index (BMI) in kg/m^2, a key indicator of healthy weight that can help identify potential health risks.
Valsalva ratio | one year
  The Valsalva ratio is the proportion of the highest and lowest heart rate during and immediately after performing a Valsalva maneuver. A value of 1.21 or more is defined as a normal response
Stand 30:15 ratio | one year
  The Stand 30:15 ratio is the ratio of the highest heart rate during (occurring approximately 15 sec after the initiation of standing) and immediately following standing up from a supine position (occurring approximately 30 sec after the initiation of standing).
deep breath test interpretation | one year
  The heart rate response to deep breathing test was calculated as the difference between maximum heart rate during inhalation and minimum heart rate during exhalation.
  A difference of 15 beats/min or more is considered parasympathetic activation.

SECONDARY OUTCOMES:
Framingham risk score (FRS) | one year
  The Framingham risk score predicts cardiovascular disease risk in asymptomatic patients. The risk is considered low if Framingham Risk Score is less than 10%, moderate if it is 10% to 19%, and high if it is higher than 20%. Heart rate variability (HRV) may be correlated with the Framingham risk score when analyzing the effects of different anti-diabetic drugs. It is expected that if the Heart Rate Variability decreases, the Framingham score will increase, indicating a higher risk of Atherosclerotic Cardiovascular disease risk in the next 10 years. Conversely, if Heart Rate Variability increases, the Framingham score may decrease, indicating a reduced risk of Atherosclerotic cardiovascular disease risk.

CONTACTS AND LOCATIONS:
Overall Officials: Labiba K. El-Khordagui, Prof. Dr., Study Director — Alexandria University; Ahmed F. El-Yazbi, Prof. Dr., Study Director — Alamein International University and Alexandria University; Mohamed I. Sanhoury, Ass. prof., Study Director — Alexandria University
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] American Diabetes Association Professional Practice Committee. 2. Diagnosis and Classification of Diabetes: Standards of Care in Diabetes-2024. Diabetes Care. 2024 Jan 1;47(Suppl 1):S20-S42. doi: 10.2337/dc24-S002. PMID 38078589
- [Result] Risk M, Bril V, Broadbridge C, Cohen A. Heart rate variability measurement in diabetic neuropathy: review of methods. Diabetes Technol Ther. 2001 Spring;3(1):63-76. doi: 10.1089/152091501750220028. PMID 11469709
- [Result] Bosomworth NJ. Practical use of the Framingham risk score in primary prevention: Canadian perspective. Can Fam Physician. 2011 Apr;57(4):417-23. PMID 21626897